CLINICAL TRIAL: NCT03643393
Title: Report 2 Cases of Massive Incarceration Necrosis Rectal Prolapse Are Successfully Treated With Altemeier's Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viet Duc University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMTT-VD-2018
Record Dates: First submitted 2018-07-31; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- incarceration rectal prolapse (Other)
  Interventions: Procedure: perineal rectosigmoidectomy

INTERVENTIONS:
Procedure: perineal rectosigmoidectomy — In an Altemeier perineal rectosigmoidectomy, a full-thickness circumferential incision is made in the prolapsed rectum about 1-2 cm from the dentate line (see the image below). The hernia sac is entered, and the prolapse is delivered. The mesentery of the prolapsed bowel is serially ligated until no further redundant bowel can be pulled down. The bowel is transected and either hand-sewn to the distal anal canal or stapled with a circular stapler. Before anastomosis, some surgeons plicate the levator ani muscles anteriorly, which may help improve continence.
  Other Names: Altemeier's procedure

SUMMARY:
Incarceration and necrosis of rectal prolapse is rare and often requires urgent management. Perineal rectosigmoidectomy (Altemeir procedure) is a reasonable technique for this condition. The need for a diverting stoma depends on the patient's condition and the experience and judgement of the surgeon. A literature review was performed to determine optimal management of incarcerated and necrotic rectal prolapse, and to determine the indication for fecal diversion.

ELIGIBILITY:
Inclusion Criteria:

* 2 cases incarceration rectalprolapse

Exclusion Criteria:

* N/A

Ages: 52 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
recurrent rectal prolapse | 3 months after surgery
  patients were asked for symptoms such as: pain during bowel movements, mucus or blood discharge from the protruding tissue, a loss of urge to defecate, awareness of something protruding upon wiping

CONTACTS AND LOCATIONS:
Overall Officials: xuan hung nguyen, DR, Study Chair — center of colorectal surgery - viet duc university hospital

IPD SHARING:
Plan to Share IPD: Undecided